CLINICAL TRIAL: NCT00321295
Title: Prospective Evaluation Of Biventricular Pacing In Patients With Left Ventricular Dysfunction After Cardiovascular Surgery
Brief Title: Biventricular Pacing In Patients With Left Ventricular Dysfunction After Cardiovascular Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Haines, David MD (Unknown)
Responsible Party: Evonich, MD, Rudolph, William Beaumont Hospitals
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HIC 2004-083
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Cardiomyopathy; Heart Failure, Congestive; Thoracic Surgery
Keywords: Bi-ventricular pacing; Cardiac Surgery; Cardiomyopahty; Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure

INTERVENTIONS:
Device: Atrial synchronous bi-ventricular pacing

SUMMARY:
Congestive heart failure (CHF) is a medical condition that is due to left ventricular systolic dysfunction (LVSD). LVSD is a decreased ability of the heart to pump blood forward. There are 5 million people in the United States that have CHF and 52,828 new cases are diagnosed annually. There are 995,000 hospital visits and 52,828 deaths annually due to CHF. Previous studies have shown that people with this condition are at a higher risk for complications immediately after any type of heart surgery than are normal individuals. This includes increased dependence on medications and devices to improve the pumping function of the heart and blood pressure. Additionally, they also have longer lengths of hospital stay and higher rates of death compared to normal individuals.

Some patients with LVSD not only have a decreased pumping ability of the heart, they also have an inefficient pumping function. These patients have been shown to benefit from a device therapy known as biventricular pacing. Biventricular pacing involves simultaneously electrically stimulating the two major pumping chambers of the heart known as ventricles using a pacemaker and wires. This causes a more coordinated contraction of the heart chambers resulting in improvement in the pumping ability of the heart and blood pressure. Studies have confirmed that in these patients, implantation of a biventricular pacemaker improves patients' symptoms and quality of life as well as decreasing a need for future hospitalizations. Whether biventricular pacing in patients with LVSD improves patient outcomes after heart surgery has not been investigated.

Some patients temporarily develop slow heart rates after cardiovascular surgery. These slow heart rates can cause a decrease in the blood pumped from the heart and result in low blood pressures. Therefore, all patients undergoing cardiovascular surgery, regardless of left ventricular function, receive temporary pacing wires that are placed on one of the ventricles during the surgery. Temporary pacing will result in an increase in heart rate and improvement in the amount of blood pumped by the heart and in blood pressure. The placement of these wires is precautionary as only a few patients need to be paced for slow heart rates. Once patients are felt to no longer require them, the wires are easily removed. The purpose of this study is to determine whether biventricular pacing immediately after heart surgery in patients with LVSD will improve in-hospital outcomes.

Patients that are scheduled for heart surgery and meet the inclusion criteria will be approached for consent to participate in this study. Once consented, they will be randomized to one of three treatment arms: usual care, RV pacing (single ventricle pacing), or biventricular pacing. Randomization is a process similar to picking numbers out of a hat. The patients will then undergo surgery as scheduled. During the surgery, the patients will receive the temporary pacing wires on both ventricles instead of one. Immediately after surgery, the patients will receive either usual care, RV pacing, or biventricular pacing depending upon the treatment arm that they were randomized to. The pacing wires will be removed as soon as the patients become stable as per routine. The clinical, operative, and in-hospital characteristics of these patients will be recorded on specialized forms. The characteristics of those that received biventricular pacing will be compared to those that had RV or no pacing to see whether there was any benefit to this mode of therapy.

DETAILED DESCRIPTION:
1. Basis for the study/study rationale Patients with congestive heart failure have high rates of mortality and morbidity (1). There are 5 million people in the United States that have congestive heart failure (CHF) and 52,828 new cases are diagnosed annually. There are 995,000 hospital visits with 52,828 deaths annually due to this condition. Although there have been numerous medical advances in drug therapy, there was a 164% increase in the number of hospital admissions for CHF since 1979 (1, 2).

   Biventricular (BiV) pacing has been shown to have acute and chronic benefits in a subset of patients with CHF (3-6). Those that have been shown to benefit from this mode of therapy have left ventricular systolic dysfunction with a widened QRS duration on the electrocardiogram. Acute hemodynamic studies comparing patients at baseline with either right ventricular (RV) or BiV pacing show significant improvements in the systolic blood pressure and cardiac output in patients with BiV pacing compared to either RV pacing or baseline measurements (3, 4). Furthermore, BiV pacing was associated with decrease in the pulmonary capillary wedge pressure (PCWP) and diastolic mitral regurgitation. These acute hemodynamic benefits are sustained and manifest as improvements in clinical symptoms. The Multisite Stimulation in Cardiomyopathies (MUSTIC) study showed that BiV pacing was associated with a 23% increase in the distance walked in six minutes (P<0.001), a 32% increase in the quality-of-life score (P<0.001), an 8% increase in the peak oxygen uptake (P<0.03), and a 66% decrease in the need for hospitalization (P<0.05) compared to no pacing (5). Patients also preferred BiV pacing compared to no pacing (P<0.001). The Multicenter InSync Randomized Clinical Evaluation (MIRACLE) study not only confirmed many of the findings of the MUSTIC trial, but also showed improvement in the left ventricular ejection fraction (LVEF) with BiV pacing (+4.6% vs. -0.2%, P<0.001), compared to non-paced controls (6). Such data has led to the classification of BiV pacing in patients with dilated cardiomyopathy as a class IIa recommendation by ACC/AHA/NASPE guidelines (7).

   Coronary artery bypass grafting (CABG) in patients with left ventricular dysfunction carries a high mortality (8). Furthermore, patients with a low LVEF have a greater need for intraaortic balloon pump (P<0.0001) and inotropic support (P<0.001) with a longer length of hospital stay (P<0.002) compared with those with normal LVEF (9, 10).

   Conduction system abnormalities following CABG are common (11, 12). The majority of these abnormalities are transient and are often managed using temporary epicardial pacing. Hence, all patients that undergo CABG receive epicardial leads as a precautionary measure. These leads are placed on the right or left ventricle and the right atrium. When patients are felt to no longer require these, they are removed easily. The role of BiV pacing in this setting is unknown. Whether patients that have left ventricular dysfunction would have improved post-operative mortality, less need for intraaortic balloon pump and inotropic support, and shorter length of hospital stay is unknown.
2. Objectives Our hypothesis is that BiV pacing immediately following CABG will improve in-hospital outcomes in patients with left ventricular systolic dysfunction.

   Endpoints:

   Primary: -Length of ICU stay

   Secondary: -In-hospital mortality
   * Length of hospital stay
   * Duration of inotropic support
   * Duration of intraaortic ballon pump support
   * Duration of mechanical ventillation
   * Change in stroke volume with biventricular pacing
   * Change in ventricular synchrony with biventricular pacing
3. Methodology All patients that are scheduled for CABG or valve surgery and meet the inclusion criteria will be approached for consent pre-operatively. Once consent is obtained the patient will be randomized into one of three treatment arms: usual care, RV pacing, or BiV pacing. The patients will then undergo surgery as per routine. During cardiovascular surgery patients routinely receive epicardial pacing leads that are placed on the right or left ventricle and the right atrium. For the purposes of this study, epicardial pacing leads will be placed on both the right and left ventricles as well as the right atrium.

   After surgery is completed, the patients will receive either usual care, RV pacing, or BiV pacing depending upon their treatment arms. Intraoperative transesophageal echocardiography (TEE) is routinely performed during cardiac surgery. If TEE is being used in the subject images will be recorded with biventricular pacing, right ventricular pacing and no pacing in the first 30 patients studied to quantify changes in vetricular synchrony with biventricular pacing. Once the patient arrives in the SICU hemodynmic monitoring will be performed as usual. All patients return from the operating room with a pulmonary artery catheter. In the first 50 patients the stroke volume will be obtained by thermodilution method using the pulmonary artery catheter in their assigned treatment arm as well as following 2 minutes of right ventricular pacing and again following 2 minutes of biventricular pacing. Pacing will be continued in the assigned treatment arm until all inotropic and intraortic ballon pump support has been weaned off. Crossover in treatment arms is discouraged, but will be at the discretion of the treating physicians. The epicardial pacing leads will be removed as per routine.
4. Inclusion/Exclusion Criteria

   Inclusion Criteria:
   1. Age > 18 years
   2. Planned CABG and/or valve surgery
   3. LVEF < 30%
   4. Able to give written informed consent

   Exclusion Criteria:
   1. Enrollment in other research protocols
   2. Inability to give written informed consent
   3. Pregnancy
5. Methods of data acquisition and analysis Clinical, operative, and in-hospital information for each subject will be recorded on standardized case report forms (see attached) at the time of hospitalization or soon after discharge. The characteristics of those that received BiV pacing will be compared to those that received either no pacing or RV pacing. The data will be recorded in a manner such that there are no patient identifiers. The information will then be transferred to a computer database. The case report forms will be kept under lock and key on the third floor of the WBH Heart Center. The computer data base will be password protected. Only the investigators will have access to the case report forms or computer database.
6. References

   1. American Heart Association. Heart Disease and Stroke Statistics - 2004Update. Dallas, Texas: American Heart Association; 2003.
   2. Braunwald E, Bristow MR. Congestive heart failure: fifty years of progress. Circulation 2000; 102 (suppl 4):IV14-IV23.
   3. Blanc JJ, Etienne Y, Gilard M et al. Evaluation of different ventricular pacing sites in patients with severe heart failure. Results of an acute hemodynamic study. Circulation 1997;96:3273-3277.
   4. Leclercq C, Cazeau S, Breton HL et al. Acute hemodynamic effects of biventricular DDD pacing in patients with end-stage heart failure. J Am Coll Cardiol 1998;32:1825-1831.
   5. Cazeau S, Leclercq C, Lavergne T et al. Effects of multisite biventricular pacing in patients with heart failure and intraventricular conduction delay. N Engl J Med 2001;334:873-80.
   6. Abraham WT, Fisher WG, Smith AL et al. Cardiac resynchronization in chronic heart failure. N Engl J Med 2002;346:1845-53.
   7. Gregoratos G, Abrams J, Epstein AE et al. ACC/AHA/NASPE 2002 guideline update for implantation of cardiac pacemakers and antiarrhythmia devices: summary article: a report of the Am College of Cardiology/Am Heart Association Task Force on Practice Guidelines (ACC/AHA/NASPE Committee to Update the 1998 Pacemaker Guidelines). Circulation 2002;106:2145-2161.
   8. Alderman EL, Fisher LD, Litwin P et al. Results of coronary artery surgery in patients with poor left ventricular function (CASS). Circulation 1983;68:785-95.
   9. Trachiotis GD, Weintraub WS, Johnston TS et al. Coronary artery bypass grafting in patients with advanced left ventricular dysfunction. Ann Thorac Surg 1998;66:1632-1639.
   10. Antunes PE, Ferrao de Oliveira JM, and Antunes MJ. Coronary surgery with non-cardioplegic methods in patients with advanced left ventricular dysfunction: immediate and long term results. Heart 2003;89:427-431.
   11. Pires LA, Wagshal AB, Lancey R et al. Arrhythmias and conduction disturbances after coronary artery bypass graft surgery: epidemiology, management, and prognosis. Am Heart J 1995;129:799-808.
   12. Mustonen P, Hippelainen M, Vanninen E et al. Significance of coronary artery bypass grafting-associated conduction defects. Am J Cardiol 1998;81:558-563.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Planned CABG and/or valve surgery
* LVEF < 30%
* Able to give written informed consent

Exclusion Criteria:

* Enrollment in other research protocols
* Inability to give written informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Length of ICU stay

SECONDARY OUTCOMES:
In-hospital mortality
Length of hospital stay
Duration of inotropic support
Duration of intraaortic ballon pump support
Duration of mechanical ventillation
Change in stroke volume with biventricular pacing
Change in ventricular synchrony with biventricular pacing

CONTACTS AND LOCATIONS:
Overall Officials: Rudolph F Evonich, MD, Principal Investigator — Corewell Health East; David E Haines, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States